CLINICAL TRIAL: NCT05523427
Title: Two Lactobacilli Strains as Adjuvant Therapy in the Management of Irritable Bowel Syndrome: A Randomized Clinical Trial
Brief Title: Probiotics as Adjuvant Therapy in the Management of Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mosul (Other)
Responsible Party: Principal Investigator, Radhwan Al-Zidan, Lecturer, University of Mosul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCMRE-phA-22-11
Record Dates: First submitted 2022-08-29; First posted 2022-08-31 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Irritable Bowel Syndrome; Irritable Bowel Syndrome With Diarrhea
Keywords: IBS; IBS-D; Abdominal pain; Abdominal distention; Probiotic; Lactobacilli; Mucus; L. plantarum; L. acidophilus
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment of IBS (No Intervention): Mebeverine 135 mg Sulpiride 25 mg Simethicone 200 mg
  They were administered in a single capsule, three time daily before meals.
- Probiotics + Standard treatment of IBS (Experimental): A capsule containing the L. plantarum and L. acidophilus strains is to be administered twice daily for three months in addition to the standard treatment of IBS.
  Interventions: Dietary Supplement: Two probiotic strains (L. plantarum and L. acidophilus)

INTERVENTIONS:
Dietary Supplement: Two probiotic strains (L. plantarum and L. acidophilus) — A capsule containing the L. plantarum and L. acidophilus strains is to be administered twice daily for three months in addition to the standard treatment of IBS.
  Arms: Probiotics + Standard treatment of IBS

SUMMARY:
Studying the effects of adding probiotics to the drug regimen of patients with diarrhea predominant IBS

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a common highly prevalent functional gastrointestinal (GI) disorder that places an enormous burden on resource-challenged healthcare systems. Although many drugs have been advocated in the treatment of IBS, including psychotropic agents, antispasmodics, bulking agents, and 5-HT receptor antagonists. However, in the vast majority of instances, these medications have failed to provide adequate symptom alleviation, presumably due to the disease's diverse pathophysiology. Probiotics are "live bacteria that confer a health benefit on the host when administered in suitable doses". In IBS, a decrease in Bifidobacterium and Lactobacillus species, as well as an increase in Gamma-proteobacteria species (a family of pathogens), has been described in IBS studies. Therefore, the ability of probiotics to repair dysbiosis (qualitative and quantitative changes in the microbiota) or stabilize the host microbiota is the reason for their use in the treatment of IBS.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16-55
2. Both genders
3. Patients diagnosed clinically with IBS based on Rome's criteria
4. IBS-Diarrhea only with pain & distention
5. Duration of symptoms 6 months

Exclusion Criteria:

1. Age > 55
2. Celiac disease
3. Inflammatory bowel disease (ulcerative colitis & Crohn's)
4. Thyroid disease
5. Colonic CA
6. Lactose intolerance
7. Alarming features (anemia, blood in the stool, weight loss, abdominal masses, dysphagia, family history of GIT malignancy)
8. Preexisting use of antibiotics in the previous 3 months.
9. Preexisting systemic diseases

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
The change in bowel habits (based on the IBS-SSS) after treatment with a multi-strain probiotic or standard treatment, and compared with baseline. | Three months
  The change in severity of abdominal pain and distention, frequency of bowel motion, satisfaction with bowel habits, and IBS-related quality of life (QoL).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Mosul, Mosul, Ninevah, Iraq

IPD SHARING:
Plan to Share IPD: No